CLINICAL TRIAL: NCT04426487
Title: Effect of Progesterone Therapy in Cases With Traumatic Subarachinoid Haemorrhage on Clinical Outcome and Resistive Vasculer Indices of Middle Cerebral Artery Transcranial Doppler
Brief Title: Effect of Progesterone Therapy on Traumatic Subarachinoid Haemorrhage on Clinical Outcome and Resistive Vasculer Indices of Middle Cerebral Artery Transcranial Doppler
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Principle investigator, Ministry of Health and Population, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 625/4-2020
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Traumatic Brain Injury
Keywords: Progesterone; Transcranial doppler
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Progesterone

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): Receiving conventional management for traumatic subarachinoid hemorrhage
  Interventions: Drug: Progesterone
- progesterone group (Active Comparator): Intramusculer progesterone therapy before and after craniotomy
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — Intramusculer progesterone

SUMMARY:
Traumatic subarachinoid hemorrhage is associated with serious complications related to mortality . Delayed neuronal ischemia and rebleeding are most common and serious. Progesterone can delay both .

DETAILED DESCRIPTION:
Progesterone is an neurosteroid that can help integrity of blood brain barrier . Traumatic subarachinoid hemorrhage disrupts this blood brain barrier facilitating post traumatic vasospasm and neuronal ischemia. Transcranial doppler can detect cerebral vasoconstriction through resistive vasculer indices

ELIGIBILITY:
Inclusion Criteria:

* Traumatic subarachinoid hemorrhage

Exclusion Criteria:

* History of malignency

  * History of cerebrovasculer stroke
  * Morbid obese

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-20 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants suffering neuronal infarction | 2 months
  Transcranial doppler

CONTACTS AND LOCATIONS:
Overall Officials: Hany Mikhail, MD, Study Director — Faculty of medicine. ElMinia University
Locations (1):
- ElMinia University, Minya, Abohelal, Egypt

IPD SHARING:
Plan to Share IPD: No